CLINICAL TRIAL: NCT05885230
Title: The Efficacy of Ultrasound-guided Pecto-Intercostal Fascial Plain Block Versus Lidocaine Infusion on Acute and Chronic Post-thoracotomy Pain; A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Ultrasound Guided PIFB Versus Lidocaine Infusion on Postoperative Pain After Thoracotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariana Soliman, Lecturer of anaesthesia, surgical intensive care and pain managment, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMBSUREC/09042023/Mikhael
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIFB group (Active Comparator): patients will receive bilateral ultrasound-guided pecto-intercostal fascial block using 20 ml of bupivacaine 0.25% for each side.
  Interventions: Procedure: pecto intercostal fascial block using bupivacaine 0.25%
- LIDOCAINE group (Active Comparator): 1.5 mg/kg lidocaine will be administered after induction of anesthesia, then 2mg/kg/h lidocaine will be administered with continuous intravenous infusion until the end of the surgery.
  Interventions: Drug: lidocaine infusion

INTERVENTIONS:
Procedure: pecto intercostal fascial block using bupivacaine 0.25% — patients will receive bilateral ultrasound-guided pecto-intercostal fascial block using 20 ml of bupivacaine 0.25% for each side.
  Other Names: Sunnypivacaine
  Arms: PIFB group
Drug: lidocaine infusion — 1.5 mg/kg lidocaine will be administered after induction of anesthesia, then 2mg/kg/h lidocaine will be administered with continuous intravenous infusion until the end of the surgery.
  Other Names: Lignocaine
  Arms: LIDOCAINE group

SUMMARY:
Chronic pain is a common complication after cardiothoracic surgery. The prevalence of post-thoracotomy pain syndrome (PTPS) ranges from 33% to 91%. Exact pathogenetic mechanisms for developing chronic pain after thoracotomy are unknown. Apart from intraoperative nerve damage and subsequent postoperative neuropathic pain, operation techniques, age, sex, pre-existing pain, genetic and psychosocial factors, severe postoperative pain, and analgesic management are suspected to have an impact on the development of PTPS .

DETAILED DESCRIPTION:
Ultrasound-guided Pecto-intercostal Fascial Block (PIFB) has been advocated by some researchers for cardiac surgery. Pecto-intercostal fascial plane block (PIFB) is a novel, minimally invasive, regional fascial plane block technique. PIFB was first described by de la Torre in patients undergoing breast surgery . PIFB targets the anterior intercostal nerves as they run in the fascial plane between the pectoral and the intercostal muscles and emerge on either side of the sternum.

Also, lidocaine, a short-acting local anesthetic, has been proved to have analgesic and anti-inflammatory effects . The application of lidocaine by continuous infusion in the intraoperative period and immediately after the surgery appears to reduce the immediate postoperative pain, and may prevent the PTPS

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years.
2. patient scheduled to undergo elective on-pump cardiac surgery with sternotomy.
3. American Society of Anesthesiologists classification of physical status < IV.

Exclusion Criteria:

1. emergency surgery.
2. off-pump surgery.
3. redo surgery.
4. ejection fraction less than 35%.
5. refusal of the patient.
6. known hypersensitivity to LA.
7. chronic opioid use or chronic pain patient.
8. psychiatric problems or communication difficulties.
9. liver insufficiency (defined as a serum bilirubin ≥ 34 μmol/l, albumin ≤ 35 g/dl, INR ≥ 1.7).
10. renal insufficiency (defined as a glomerular filtration rate < 44 ml/min).
11. obstructive sleep apnea syndrom.
12. coexisting hematologic disorders.
13. pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Total dose of morphine in the first 24 h postoperatively. | 24 hours postoperative
  total morphine consumed in the first 24 hour

SECONDARY OUTCOMES:
NRS numerical rating scale. | 24 hours post operative
  NRS ranging from grade 0 (no pain) to grade 10 (most severe pain) NRS< 4 is acceptable for pain relief
chronic postoperative pain in 3 months after operation according to numerical rating scale | within 3 months postoperative
  NRS ranging from grade 0 (no pain) to grade 10 (most severe pain) NRS< 4 is acceptable for pain relief
Time to rescue analgesic | within 24 hour postoperative
  time from extubation to the time the patiants given analgesia
time to extubation | within 24 hour post operative
  from end of surgery to the time of extubation
length of intensive care stay | within one week
  from end of surgery to the time of discharging to the surgical word

CONTACTS AND LOCATIONS:
Overall Officials: Mariana A mansour, Lecturer, Principal Investigator — benisuef university hospital,Egypt
Locations (1):
- Benisuef University Hospital, Banī Suwayf, e\EYGPT, Egypt